CLINICAL TRIAL: NCT00835445
Title: Nasal Features of Subjects With Nasal Polyposis With or Without Asthma
Brief Title: Biopsies and Polyps
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Louis-Philippe Boulet, Hôpital Laval
Other Study IDs: CER 20188
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2010-12

CONDITIONS: Nasal Polyps; Asthma
MeSH Terms: conditions — Nasal Polyps; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal polyps (Biopsies) Normal nasal mucosa (Biopsies) Sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Asthmatics with polyps
- 2: Non-asthmatics with polyps

SUMMARY:
Background: Nasal polyps are found in about 5% of asthmatic patients.A close link exists between the upper and lower airways and the concept of the "United Airways" has emerged mainly from studies on allergic rhinitis and asthma. However, other upper airway diseases, such as chronic sinusitis and nasal polyposis may influence lower airway diseases. As for nasal polyposis, eosinophils are the major effector cells in asthma and have been associated with a worsening of this condition.

Aim: To compare normal nasal mucosa and nasal polyp biopsies from subjects with nasal polyposis with or without asthma.

Hypothesis: Nasal polyps from asthmatic subjects show a more aggressive pro-inflammatory pattern of cytokine expression compared to nasal polyps from non asthmatic subjects, and therefore contribute to the development and severity of asthma.

DETAILED DESCRIPTION:
The study will include 2 visits separated by a maximum of 7 days. During the first visit, subjects' characteristics will be documented by a locally validated questionnaire. Allergy skin prick tests, spirometry, methacholine inhalation test and induced sputum will also be done. Asthma and rhinitis control will be evaluated by locally validated questionnaires, the Asthma Control Scoring System (ACSS) and the Rhinitis Control Scoring System (RCSS), respectively. Nasal peak inspiratory flow (NPIF) and oral peak expiratory flow (PEF) will also be recorded to obtain the nasal blockage index (NBI). On the second visit, nasal biopsies will be taken.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Non smoking men or women aged 18 to 65 years old.
* Subjects will have nasal polyps as defined above.

For asthmatic subjects:

* Subjects will have a history consistent with asthma according to the criteria of the ATS[18] defined on the basis of episodic or persistent chest tightness, wheeze or cough in the past 6 months. At entry into the study, FEV1 will be over 70% predicted.
* Asthma will have been stable for at least 3 months before entering the trial.
* Asthma medication will have been stable for at least 1 month prior to the study.

For non asthmatic subjects:

* A methacholine challenge test with a PC20 (provoking concentration of methacholine to cause a 20% fall in FEV1) over 16 mg/mL.

Exclusion Criteria:

For all subjects:

* Smoking (current smoking) or ex-smoking (les than 6 months or history of more than 10 pack-year of smoking).
* Use of anti-leukotriene medication within the last 3 months.
* Use of systemic corticosteroids within the last 3 months.
* Use of anti-coagulant therapy.
* Recent (less than 1 month) upper or lower respiratory tract infection, any other condition that may interfere with the evaluations.
* Pregnancy, breast-feeding or planned pregnancy during the study. Fertile woman not using acceptable contraceptive measures, as judged by the investigator.
* Subjects unable to perform or with contraindications to the tests proposed.
* Subjects who are, in the opinion of the investigator, mentally or legally incapacitated thus preventing informed consent from being obtained.

For asthmatic subjects:

* Unstable asthma shown by respiratory symptoms and B2-agonists need more than 3 times/week and nocturnal asthma symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruited from the ENT clinic (Laval Hospital, Quebec City, Canada)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the difference in expression of IL-5 in nasal polyps and normal mucosa biopsies from asthmatic and non asthmatic subjects. | No time frame

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Centre de recherche, Hôpital Laval
Locations (1):
- Hopital Laval, Ste-Foy, Quebec, Canada